CLINICAL TRIAL: NCT06341283
Title: A Retrospective Real-world Study of Efficacy, Safety, and Economic Assessment of Abemaciclib Tablets Based on Hospital Information System(HIS) in Hormone Recepter Positive(HR+) Breast Cancer Patients
Brief Title: A Retrospective Real-world Study of Abemaciclib in HR+ Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Other Study IDs: BCOOS2024
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; Neoplasms; Breast Diseases
Keywords: Abemaciclib; Real world study; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Breast Diseases | interventions — abemaciclib; Letrozole; Anastrozole; Fulvestrant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- BCOOS-A1: The patients in this array are treated with Abemaciclib and Letrozole/Anastrozole.
  Interventions: Drug: Abemaciclib and Letrozole/Anastrozole
- BCOOS-A2: The patients in this array are treated with Letrozole or Anastrozole.
  Interventions: Drug: Letrozole or Anastrozole
- BCOOS-B1: The patients in this array are treated with Abemaciclib and Fulvestrant.
  Interventions: Drug: Abemaciclib and Fulvestrant
- BCOOS-B2: The patients in this array are treated with Fulvestrant only.
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Abemaciclib and Letrozole/Anastrozole — Take the treatment with Abemaciclib and Letrozole/Anastrozole at the same time.
  Other Names: BCOOS-A1
  Groups: BCOOS-A1
Drug: Letrozole or Anastrozole — Take the treatment with Letrozole or Anastrozole.
  Other Names: BCOOS-A2
  Groups: BCOOS-A2
Drug: Abemaciclib and Fulvestrant — Take the treatment with Abemaciclib and Fulvestrant at the same time.
  Other Names: BCOOS-B1
  Groups: BCOOS-B1
Drug: Fulvestrant — Take the treatment with Fulvestrant only.
  Other Names: BCOOS-B2
  Groups: BCOOS-B2

SUMMARY:
The present study will assess real-world clinical outcomes, adverse events and economics from treatment with endocrine therapy(ET) combined with abemaciclib in patients with hormone receptor-positive(HR+) breast cancer.

DETAILED DESCRIPTION:
Based on clinical trials data, Abemaciclib has been approved for early and advanced breast cancer with HR+ and human epidermal growth factor 2 receptor-negative(HER2-), but clinical trials require real-world research data as supplementary validation supporting evidence. This study will assess real-world clinical outcomes, adverse events and economics from treatment with endocrine therapy(ET) combined with abemaciclib in patients with HR+ breast cancer. In addition, this trial will explore the efficacy of Abemaciclib in patients with HR+ and human epidermal growth factor 2 receptor-positive(Her2+) breast cancer.

This study will now include real-world data on efficacy, toxicity and economics of abemaciclib in the adjuvant setting in HR+ breast cancer. Participants to be enrolled will come from an online platform for researches which all the privacy information has been controlled. The investigators are going to gather 2 groups of breast-cancer-one-other-study(BCOOS) including BCOOS-A and BCOOS-B. Group BCOOS-A includes the patients treated with Abemaciclib and Letrozole/Anastrozole compared with treated with Letrozole/Anastrozole only. Group BCOOS-B includes the patients treated with Abemaciclib and Fulvestrant compared with treated with Fulvestrant only.

Investigators will measure clinical outcomes, adverse events and economics in each group above.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Histologically confirmed HR-positive breast cancer and Imaging/pathological evidence of metastasis is available
* Treatment with abemaciclib in combination with endocrine therapy
* Any endocrine therapy
* Having solid tumor efficacy evaluation criteria RECIST 1.1 measurable lesions

Exclusion Criteria:

* Combined with other primary malignancies
* Associated with serious non-tumor related diseases, such as cardiovascular system, respiratory system, nervous system, blood system, digestive system
* Pregnant or lactating women
* male breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed HR-positive breast cancer treated with abemaciclib in combination with endocrine therapy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | Through the completion of the study, for an average of 6 months
  The time from treatment initiation to either the first documented disease progression or death from any cause.

SECONDARY OUTCOMES:
Objective Remission Rate(ORR) | Up to 36 months
  The proportion of patients who achieved pre-defined tumor volume reduction and maintained the minimum time limit was the sum of complete response (CR) and partial response (PR) proportions.
Disease Control Rate(DCR) | Up to 36 months
  The number of patients who achieved complete response(CR),partial response (PR) and stable lesion (SD) after treatment as a percentage of the evaluable cases
Toxicity rate | Up to 36 months
  Adverse events from the time from treatment initiation to disease progression, patient death or last recorded
Cost-utility analysis(CUA) | Up to 36 months
  In health economics the purpose of CUA is to estimate the ratio between the cost of a health-related intervention and the benefit it produces in terms of the number of years lived in full health by the beneficiaries.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cao, docter, Study Director — The Affiliated Hospital of Qingdao University
Locations (1):
- Clinical Research Center, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zhang QY, Sun T, Yin YM, Li HP, Yan M, Tong ZS, Oppermann CP, Liu YP, Costa R, Li M, Cheng Y, Ouyang QC, Chen X, Liao N, Wu XH, Wang XJ, Feng JF, Hegg R, Kanakasetty GB, Coccia-Portugal MA, Han RB, Lu Y, Chi HD, Jiang ZF, Hu XC. MONARCH plus: abemaciclib plus endocrine therapy in women with HR+/HER2- advanced breast cancer: the multinational randomized phase III study. Ther Adv Med Oncol. 2020 Oct 22;12:1758835920963925. doi: 10.1177/1758835920963925. eCollection 2020. PMID 33149768